CLINICAL TRIAL: NCT05155917
Title: Concurrent Subcutaneous Basal Insulin and Intravenous Insulin Pump in Hyperglycemic Crisis Patients Under Critical Care
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 210201
Record Dates: First submitted 2021-07-27; First posted 2021-12-14 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-12

CONDITIONS: Hyperglycaemic Crisis in Diabetes Mellitus; Diabetic Ketoacidosis; Hyperglycaemic Hyperosmolar Nonketotic Syndrome
Keywords: hyperglycemic crisis; DKA; HHS; insulin pump; basal insulin; critical care
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- basal insulin and insulin pump (Experimental): Subjects in the intervention group received insulin glargine sc (0.25 U/kg body weight) within 6 h of initiation of iv insulin infusion, as close to initiation of iv insulin as possible.
  Interventions: Drug: Insulin Glargine 300 UNT/ML [Toujeo]
- insulin pump (No Intervention): Patients in the control group did not receive placebo injections.

INTERVENTIONS:
Drug: Insulin Glargine 300 UNT/ML [Toujeo] — insulin glargine sc (0.25 U/kg body weight)
  Arms: basal insulin and insulin pump

SUMMARY:
The safety and efficacy of basal insulin during intravenous insulin infusion for hyperglycemic crisis patients under critical care is still unknown.

We assumed that concurrent basal insulin subcutaneous injection and intravenous insulin infusion for critically ill DKA and HHS patients would shorten the time of hyperglycemic crisis correction and achieved better glycemic control(decrease hypoglycemia and rebound hyperglycemia).

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic state (HHS) are hyperglycemic crises sharing similar clinical features including hyperglycemia, dehydration and electrolytes abnormalities. Hyperglycemia results from relative deficient circulating insulin and oversecretion of glucagon, catecholamines, cortisol, and growth hormone. Glycosuria induced osmotic diuresis leads to dehydration and electrolyte abnormalities. Diabetic ketoacidosis is also characterized by increased gluconeogenesis, lipolysis, ketogenesis, and decreased glycolysis.[1] In critically ill and mentally obtunded patients with DKA or hyperosmolar hyperglycemia, continuous intravenous insulin is the standard of care.[2] Administration of subcutaneous insulin glargine during intravenous insulin infusion shortened the time of DKA correction and significantly decreased hyperglycemia after discontinuation of the intravenous insulin. [3, 4]The differences in rebound hyperglycemia rates were highly significant for at least 12 hours after transition to subcutaneous insulin regimens in the DKA and non-DKA patients as well as in organ transplant patients receiving steroids. [4] However, the previous studies only enrolled small numbers of patients(without Asian population) and excluded newly diagnosed hyperglycemia or critical illness and pregnant women. The safety and efficacy of basal insulin during intravenous insulin infusion for hyperglycemic crisis patients under critical care is still unknown.

The investigators assumed that concurrent basal insulin subcutaneous injection and intravenous insulin infusion for critically ill DKA and HHS patients would shorten the time of hyperglycemic crisis correction and achieved better glycemic control(decrease hypoglycemia and rebound hyperglycemia).

ELIGIBILITY:
Inclusion Criteria:

* Patients with hyperglycemic crisis(DKA, HHS or mixing type) receiving iv insulin infusion
* Patients admitted to the Changhua Christian Hospital Medical Intensive Care Unit(MICU)

Exclusion Criteria:

* pregnancy
* age under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
the rates of rebound hyperglycemia | "the next 12 hours" after ceasing insulin infusion
  the rates of hyperglycemia( serum glucose >300mg/dl) after ceasing insulin infusion
the rates of hypoglycemia | "the next 12 hours" after ceasing insulin infusion
  the rates of hypoglycemia( serum glucose <70mg/dl) during insulin infusion

SECONDARY OUTCOMES:
insulin infusion time | 'the next 12 hours' after ceasing insulin infusion
  hours of the total insulin infusion therapeutic time
ICU length of stay | through study completion, an average of 1 year
  days of ICU admission
ventilator use days | through study completion, an average of 1 year
  days of ventilator depending time(from intubation to extubation)
ICU Mortality rate | through study completion, an average of 1 year
  mortality rate during ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dhatariya K, Mustafa O, Stathi D. Hyperglycemic Crises. 2025 Jun 10. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK279052/ PMID 25905280
- [Result] American Diabetes Association. 15. Diabetes Care in the Hospital: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S193-S202. doi: 10.2337/dc20-S015. PMID 31862758
- [Result] Shankar V, Haque A, Churchwell KB, Russell W. Insulin glargine supplementation during early management phase of diabetic ketoacidosis in children. Intensive Care Med. 2007 Jul;33(7):1173-1178. doi: 10.1007/s00134-007-0674-3. Epub 2007 May 17. PMID 17508198
- [Result] Hsia E, Seggelke S, Gibbs J, Hawkins RM, Cohlmia E, Rasouli N, Wang C, Kam I, Draznin B. Subcutaneous administration of glargine to diabetic patients receiving insulin infusion prevents rebound hyperglycemia. J Clin Endocrinol Metab. 2012 Sep;97(9):3132-7. doi: 10.1210/jc.2012-1244. Epub 2012 Jun 8. PMID 22685233